CLINICAL TRIAL: NCT02700776
Title: 1380GCC: Prospective Study of GP-88 Blood Test in Healthy Women With Baseline Gail Model Risk Assessment Undergoing Screening for Breast Cancer
Acronym: 1380GCC
Status: Terminated | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: A&G Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: HP-00058144 1380GCC
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: screening mammogram; GP88; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Measure the level of GP88 in the blood of healthy women who are having mammography screening for breast cancer. If study doctor refers subject for breast biopsy the investigator will collect the information from the biopsy.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- COHORT I-BIRADS 1 or 2,: Phlebotomy - Blood sampling for GP88 and MM. Occurs at months 0 and 6-12.
  Interventions: Other: Phlebotomy - Blood sampling for GP88 at MM
- COHORT II -BIRADS 3: Phlebotomy - Blood sampling for GP88 and MM. Occurs at months 0, 3-6, and 6-12.
  Interventions: Other: Phlebotomy - Blood sampling for GP88 at MM
- COHORT III-BIRADS 4-6: SOC Tissue Biopsy. Occurs at months 0, 3-6, and 6-12.
  Interventions: Other: Phlebotomy - Blood sampling for GP88 at MM; Procedure: SOC Tissue biopsy

INTERVENTIONS:
Other: Phlebotomy - Blood sampling for GP88 at MM — Women undergoing a screening mammogram will have a blood sample drawn to look for GP88.
  Other Names: GP88
Procedure: SOC Tissue biopsy — standard of care tissue biopsy if clinically indicated.
  Groups: COHORT III-BIRADS 4-6

SUMMARY:
The purpose of this study is find out if a protein level in the blood (called PC Cell Derived Growth Factor or glycoprotein 88 [GP88]), combined with standard mammography screening, can help detect breast cancer better than mammography screening alone. Earlier research has shown that a certain glycoprotein 88 (GP88) is higher in women with breast cancer.

In this study, investigators will measure the level of GP88 in the blood of healthy women who are having mammography screening for breast cancer. The investigator plans to correlate the results of the mammogram with the GP-88 level.

DETAILED DESCRIPTION:
Eligible healthy women >= 40 years old at average risk for developing breast cancer will be offered participation in the study at the time they present for routine screening mammogram (MM) at the University of Maryland Breast Screening Center and Baltimore Washington Medical Center; includes women who present to the center as a referral for further diagnostic workup of recent screening diagnosis of breast cancer <= to 3 months with mammographic findings on screening MM with BIRADS 0-6<= 3 months.

Informed consent will be reviewed with the study participant and She will be asked if She wishes to participate in this study. Once the volunteer agrees and signs the consent, her eligibility criteria will be reviewed by the study coordinator and if eligible the patient will be enrolled. Her MM, US or MRI results will be obtained and the study subject will be assigned to one of the 3 cohorts of patients.

COHORT I-BIRADS 1 or 2, COHORT II -BIRADS 3 COHORT III-BIRADS 4-6.

The first blood sample (20ml) for GP-88 will be drawn within 31 days of the initial signing of the informed consent. It is expected that majority of women attending the screening and diagnostic program at the UM Breast Center will be approached about this study. The investigator expects to screen 1400 and consent approximately 800 women in 12 months.

Once deemed eligible the study participant will have their first GP-88 blood sample drawn (20ml) within 31 days of signing the consent. The investigator will make every effort to draw the blood sample for GP-88 on the day of the visit to our breast center and will try not to ask study participants to come back to have the blood samples drawn unless the patient is willing to do it. However the study participant does have the option to have the GP-88 blood sample drawn within 31 days of her screening or diagnostic MM, US or breast MRI or biopsy if she wishes to participate but cannot do it on the day of her visit here. If the initial-first blood sample is never drawn the patient will be considered a screen failure, if subsequent blood samples will not be drawn or if the patient does not return for follow up screening or diagnostic MM or other testing as recommended by the radiologists, she will be replaced by another subject.

ELIGIBILITY:
Inclusion Criteria:

* Female greater than or equal to 40 years.
* Presenting to UM Breast Center and BWMC for breast imaging: screening or diagnostic mammogram, breast ultrasound (US), breast MRI, stereotactic core needle biopsy, ultrasound core needle biopsy, MRI guided breast biopsy.
* Patients with a recent screening diagnosis of breast cancer < = 3months.
* Patients presenting with mammogram findings with BIRADS of 0-6 < =3 months.
* Able to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with a personal history of stage 0-4 breast cancer >3months.
* Patients who have known severe and/or uncontrolled medical or psychiatric conditions or other conditions that could affect their participation in the study, or personal history of other malignancies.
* Patients who are unfit or unable to comply with having breast imaging studies such as mammogram, ultrasound, and MRI or breast biopsy or with study procedures-blood draw.
* Patients with personal history of ovarian cancer or other cancers.
* Patients with a personal history of breast biopsy positive for atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH), lobular carcinoma in situ (LCIS).

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prospectively determine the GP-88 blood levels in healthy female volunteers who are undergoing routine screening mammography.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Determine the GP-88 blood levels in healthy female volunteers who are undergoing routine screening mammography | 12 months
  1. To prospectively determine the GP-88 blood levels in healthy female volunteers who are undergoing routine screening mammography at the UM Breast Center, Baltimore Washington Medical Center and other local breast imaging referral centers and in patients with biopsy-confirmed breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tkaczuk, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Baltimore Washington Medical Center, Glen Burnie, Maryland